CLINICAL TRIAL: NCT04766099
Title: Impact of a Video Education Tool for the Second Stage of Labor
Brief Title: Video Education for Labor and Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Rebecca Rimsza, Clinical Fellow, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202101089
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Pregnancy Related; Educational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (No Intervention): Standard bedside coaching by labor and delivery staff
- Educational Video (Experimental): Patients will watch the provided coaching video in addition to standard bedside coaching by labor and delivery staff
  Interventions: Other: Childbirth Educational Video

INTERVENTIONS:
Other: Childbirth Educational Video — Educational video describing techniques for pushing
  Arms: Educational Video

SUMMARY:
The second stage of labor or the pushing stage can be challenging and intimidating for patients delivering for the fist time. Among women with neuraxial anesthesia pushing may not be instinctive and therefore various coaching methods are used to maximize maternal expulsive efforts and minimize pushing time. Time intensive strategies including transperineally ultrasound and bio-feedback have been employed to assist with pushing but they are difficult to implement widely. While some women may attend birthing classes or have previously been coached on pushing prior to the onset of labor, many women are unable to access classes prior to labor or do not retain what they learned in a class weeks prior to labor. Previous studies have evaluated the effect of coached pushing on the length of second stage and have indicated that coaching can decrease the second stage up to 13 minutes. In most clinical scenarios, coaching or guidance from the nurse or provider happens once the patient attains complete dilation. There are limitations to this approach as waiting to coach after a potentially long and arduous labor is suboptimal. Therefore, we propose a randomized controlled trial investigating the use of an educational video during the first stage of labor on length of the second stage.

DETAILED DESCRIPTION:
Childbirth education is critical to maternal outcomes. Receiving formal education on the birthing process sets the stage for optimal mother/baby bonding, postpartum mood, and future interactions with healthcare professionals. The American Congress of Obstetrics and Gynecology recommends patients attend birthing classes prior to labor and delivery, however previous studies found that attendance is dropping with only 56% of first-time mothers attending childbirth education classes in 2005 compared to 70% in 2001.

Multiple barriers to accessing prenatal childbirth education have been identified. Traditionally, childbirth education classes are structured as in person lectures with multiple sessions over a period of weeks and are taken prior to the onset of labor. Most childbirth education classes have accompanying costs ranging from $20-$50 for hospital classes and hundreds of dollars for private classes. Significant barriers impact patients ability to attend these classes including difficulty obtaining childcare, financial constraints, getting time off from work, and obtaining transportation. The Coronavirus pandemic has further worsened barriers to accessing childbirth education as most in-person group classes have been cancelled due to lack of funding or need for social distancing.

Most childbirth education focuses on preparation for labor and pain management in the first stage of labor neglecting the second stage. This is the stage of labor that requires the most maternal involvement and effort. Among women with epidural anesthesia pushing may not be instinctive and hence, coaching and preparation are integral to success.

The current standard of care for teaching a patient how to push is nurse-led coaching performed at the bedside immediately before the patient starts pushing. At this point, most patients are tired, anxious, and have not had enough time to process the new knowledge learned about how to push. A long or abnormal second stage is associated with adverse outcomes such as cesarean delivery, infection, and hemorrhage. Nulliparous patients are especially vulnerable to these adverse outcomes in the second stage so long as they do not feel empowered, knowledgeable, or involved in their own birth experiences.

Previous literature shows that coached pushing can decrease second stage duration up to 13 minutes. This is important as a prolonged second stage of labor is associated with maternal and neonatal morbidity including higher rates of cesarean delivery, chorioamnionitis, perineal trauma, NICU admission, neonatal sepsis, and APGAR score < 4 at 5 minutes. In most clinical scenarios, the standard of care is coaching or guidance from the nurse or provider once the patient reaches complete dilation. There are limitations to this approach as waiting to coach after a potentially long and arduous labor course is suboptimal. While physicians and nurses are qualified to coach, they may not be universally available to all patients and the quality of coaching may be impacted by volume and acuity on Labor & Delivery.

In theory, the advent of video-based education can easily be transferred to the hospital to address this issue and allows for education during labor once an epidural is placed, the patient is comfortable, and well before pushing starts. The average duration of labor and delivery in a first-time mother ranges from 14 to 20 hours. This presents an opportune window of time for video-based childbirth education to narrow gaps in childbirth education disparities and increase maternal involvement without the barriers present in the outpatient setting. The efficacy of this novel way of providing childbirth education has not been tested.

To address this quality gap, we propose a randomized trial comparing an intrapartum video education tool to standard provider-based coaching

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Over 18 year of age
* Single fetus
* Term: has completed 36 weeks of pregnancy

Exclusion Criteria:

* fetal anomalies
* Prior cesarean delivery
* contraindication to valsalva
* blind patients
* admission in the second stage of labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 161 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Length of the Second Stage of Labor | delivery
  Time from complete dilation to delivery of the fetus

SECONDARY OUTCOMES:
Labor Satisfaction Scores | 1 day ( Assessed via survey prior to discharge from the hospital)
  Labor satisfaction as measured by the Mackey Childbirth Satisfaction Rating Scale. Scores are given by patients on a scale from 1-5 with 5 being the highest and 1 being the lowest.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca R Rimsza, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodman P, Mackey MC, Tavakoli AS. Factors related to childbirth satisfaction. J Adv Nurs. 2004 Apr;46(2):212-9. doi: 10.1111/j.1365-2648.2003.02981.x. PMID 15056335
- [Background] Committee on Obstetric Practice. Committee Opinion No. 687: Approaches to Limit Intervention During Labor and Birth. Obstet Gynecol. 2017 Feb;129(2):e20-e28. doi: 10.1097/AOG.0000000000001905. PMID 28121831
- [Background] Declercq ER, Sakala C, Corry MP, Applebaum S, Herrlich A. Major Survey Findings of Listening to Mothers(SM) III: Pregnancy and Birth: Report of the Third National U.S. Survey of Women's Childbearing Experiences. J Perinat Educ. 2014 Winter;23(1):9-16. doi: 10.1891/1058-1243.23.1.9. PMID 24453463
- [Background] Lu MC, Prentice J, Yu SM, Inkelas M, Lange LO, Halfon N. Childbirth education classes: sociodemographic disparities in attendance and the association of attendance with breastfeeding initiation. Matern Child Health J. 2003 Jun;7(2):87-93. doi: 10.1023/a:1023812826136. PMID 12870624
- [Background] Simpson KR, Newman G, Chirino OR. Patients' perspectives on the role of prepared childbirth education in decision making regarding elective labor induction. J Perinat Educ. 2010 Summer;19(3):21-32. doi: 10.1624/105812410X514396. PMID 21629391
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Fenwick J, Toohill J, Gamble J, Creedy DK, Buist A, Turkstra E, Sneddon A, Scuffham PA, Ryding EL. Effects of a midwife psycho-education intervention to reduce childbirth fear on women's birth outcomes and postpartum psychological wellbeing. BMC Pregnancy Childbirth. 2015 Oct 30;15:284. doi: 10.1186/s12884-015-0721-y. PMID 26518597
- [Background] Cankaya S, Simsek B. Effects of Antenatal Education on Fear of Birth, Depression, Anxiety, Childbirth Self-Efficacy, and Mode of Delivery in Primiparous Pregnant Women: A Prospective Randomized Controlled Study. Clin Nurs Res. 2021 Jul;30(6):818-829. doi: 10.1177/1054773820916984. Epub 2020 Apr 13. PMID 32281410
- [Background] Sperlich M, Gabriel C, St Vil NM. Preference, knowledge and utilization of midwives, childbirth education classes and doulas among U.S. black and white women: implications for pregnancy and childbirth outcomes. Soc Work Health Care. 2019 Nov-Dec;58(10):988-1001. doi: 10.1080/00981389.2019.1686679. Epub 2019 Nov 4. PMID 31682786
- [Derived] Rimsza RR, Perez M, Woolfolk C, Kelly JC, Carter EB, Frolova AI, Odibo AO, Raghuraman N. Video Instruction for Pushing in the Second Stage: a randomized controlled trial. Am J Obstet Gynecol. 2023 Jun;228(6):732.e1-732.e11. doi: 10.1016/j.ajog.2023.03.024. Epub 2023 Mar 20. PMID 36940771